CLINICAL TRIAL: NCT05428072
Title: Alcohol, Gut Leakiness, & Liver Disease
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Ali Keshavarzian, Principal Investigator, Rush University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ORA 09042105
Record Dates: First submitted 2022-06-16; First posted 2022-06-22 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Alcoholic Liver Disease
Keywords: intestinal permeability
MeSH Terms: conditions — Liver Diseases, Alcoholic

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- sugar test (Experimental): Participants will undergo 3 sugar tests followed by
  Interventions: Other: Sugar test; Drug: Aspirin Challenge

INTERVENTIONS:
Other: Sugar test — All participants will take two sugar tests ( sugar cocktail consisting of mannitol & lactulose) subjects within 2-3 days of the initial sugar test.
Drug: Aspirin Challenge — All participants will take a sugar test after 2 doses of aspirin, 1.3 g each given at 12 & 1 hour before the sugar drink.

SUMMARY:
The goal of this study is to investigate the role of gut leakiness in alcoholic liver disease. Gut leakiness may be the missing susceptibility factor that explains why some alcoholics develop liver disease and others don't. For this study, subjects 480 (240 male, 240 female, ages 18-80) will be recruited. Alcoholic subjects will be recruited from outpatient & inpatient alcohol detoxification units from Rush, Loyola & two halfway houses (one for women, one for men); patients with liver disease from GI/Hepatology Services at Rush, Hines VA Hosp & Loyola University; and controls from hospital staffs. All subjects will fill out a detailed questionnaire, be interviewed by the study coordinator & undergo an exam by the PI to ensure that all inclusion criteria are satisfied. All subjects will have a urine collection for tests of intestinal permeability (urinary sugars). Gut leakiness will be determined by the amount of sugars in the urine.

ELIGIBILITY:
Inclusion Criteria:

There are 4 different categories of participants that were used for recruitment:

Healthy controls

* Subjects must have a normal physical exam
* No GI complaints
* No known liver disease
* Normal liver function tests (ALT, AST, bilirubin, alkaline phosphatase, serum albumin)
* Consume no more than a moderate amount of alcohol (NIAAA definition [1 ]).
* These subjects should not be daily drinkers (< 3x / week) and should typically drink < 3 drinks per occasion.

Alcoholics

* Subjects should fulfill NIAAA criteria for at-risk drinking & alcohol abuse or dependence & DSM-IV criteria for alcoholism
* Each must have consumed alcohol regularly for at least the past 3 mos but must be sober for 3-7 day post-binge at the time of sugar test (except for group 7)
* Have a total regular heavy drinking history of at least 10 y (except for Group 6) the minimal period of time required for the development of ALD.

These are the different alcoholic groups and their specific inclusion criteria:

ALCOHOLICS WITHOUT LIVER DISEASE

* no clinical evidence of ALD on physical examination
* serum bilirubin or ALT or AST less than 1.25X normal
* sobriety must be <7 days at the time of sugar test.

ALCOHOLICS WITH LIVER DISEASE

* These subjects will have 1 of 3 possible grades of LD severity (mild, moderate, severe) & have either clinical evidence of LD (hepatomegaly, splenomegaly, and esophageal varices), or serum bilirubin or ALT or AST more than 1.5X normal.
* If liver biopsy or CT or ultrasound is available, there should be histological evidence of LD (alcoholic hepatitis or cirrhosis) or radiological evidence of LD (cirrhotic liver, splenomegaly, varices)
* Their sobriety must be <7 days at the time of the sugar test.

ALCOHOLICS WITH SHORT-TERM Drinking

* These subjects should fulfill the criteria of alcohol abuse
* have sobriety <7 days at the time of urine collection, but the duration of their heavy drinking must be <5 years
* They must not have any liver disease (negative serology) due to non-EtOH causes or clinical evidence of
* cirrhosis. Here, liver enzyme levels are not inclusion/exclusion criteria; but since the duration of EtOH abuse (<5 y) is too short for the development of cirrhosis, it is expected that none will have sustained elevated liver enzymes.

SOBER ALCOHOLICS WITH LD .

* Criteria is the same as Alcholics with liver disease but last drink was >7 days from the study enrollment.

Subjects with Non-alcoholic liver disease

* Criteria for LD are similar to those outlined for alcoholics with liver disease subjects except that drinking history should be similar to that of healthy volunteers. Subjects after liver transplant.
* These subjects must have successful liver transplantation at least 6 mos prior to the study and are on stable doses of immunosuppression for 3 mos.

Exclusion Criteria:

* Unreliable drinking history (to rule out closet drinkers or pretenders).
* Subjects must clearly fulfill the criteria either of "alcoholism" or of "on-drinker".
* Subjects with a drinking history of 5-9 years duration are excluded since this period is not short enough to preclude cirrhosis nor long enough to cause ALD in most subjects.
* Significant renal impairment (creatinine>l.2 mg/dL
* Diseases that affect GI motility such as scleroderma.
* insulin-requiring diabetes &/or uncontrolled diabetes (Hgb-Alc>8%)
* Clinically significant dehydration.
* clinically detectable ascites
* Significant peripheral edema
* Sepsis
* Clinically significant cardiac failure
* Regular daily use of medications that may affect intestinal permeability such as NSAIDS or intestinal motility (e.g. metoclopramide).
* Alcoholics positive for other markers of LD such as smooth muscle antibody, hepatitis B surface antigen, hepatitis C antibody or hemochromatosis
* Inability to sign an informed consent form
* Patients with low platelet count (<80k), uncorrectable prolonged PT (>15 sec), history of bleeding will be excluded from aspirin tests

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2003-01 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Changes in gut permeability | 3 days
  All participants will consume a sugar cocktail (lactulose & mannitol) and collect their urine. A urinary analysis was performed to measure the secretion of sugar and indicates gut permeability.
Changes in gut permeability after consuming aspirin | 1 day
  Participants will take will consume 2 doses of aspirin, 1.3 g each given at 12 & 1 h before taking a sugar test. A urinary analysis was performed to measure the secretion of sugar and indicates gut permeability.

CONTACTS AND LOCATIONS:
Locations (1):
- Ali Keshavarzian, Chicago, Illinois, United States

REFERENCES:
- [Derived] Swanson GR, Garg K, Shaikh M, Keshavarzian A. Increased Intestinal Permeability and Decreased Resiliency of the Intestinal Barrier in Alcoholic Liver Disease. Clin Transl Gastroenterol. 2024 Apr 1;15(4):e00689. doi: 10.14309/ctg.0000000000000689. PMID 38334953